CLINICAL TRIAL: NCT01170416
Title: Quantitative Measurements Comparing Body Surface Potentials During Pacemapping and Spontaneous Ventricular Tachycardia
Brief Title: Testing Objective Methods for Template Matching Ventricular Tachycardia and Pacemapping
Status: Completed | Type: Observational
Sponsor: John Sapp (Other)
Responsible Party: Sponsor-Investigator, John Sapp, Electrophysiologist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Other Study IDs: SP12
Record Dates: First submitted 2010-07-25; First posted 2010-07-27 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Ventricular Tachycardia
Keywords: Ventricular Tachycardia; Body Surface Mapping
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 12-Lead Body Surface Mapping - Focal VT .: Body surface mapping (BSM) will be completed in patients with a defined focal VT site during the EP study.
  Interventions: Other: 12-lead body surface mapping
- 12-Lead BSPM - Scar related VT, exit not identified: Body surface mapping will be competed on patients with scar related VT where the exit cannot be identified
  Interventions: Other: 12-lead body surface mapping
- 12-Lead BSPM - Scar related VT exit identified: Body surface mapping will be competed on patients with scar related VT where the exit is identified
  Interventions: Other: 12-lead body surface mapping
- 12-Lead BSPM - Supraventricular tachycardia: Body surface mapping will be completed on patients requiring an EP study for the treatment of symptoms related to supraventricular tachycardia
  Interventions: Other: 12-lead body surface mapping

INTERVENTIONS:
Other: 12-lead body surface mapping — An average of 20 distinct left ventricular sites will be mapped using 12-lead body surface mapping electrodes and recorded for 15 seconds, then sent to a computer for further analysis.

SUMMARY:
Patients sometimes suffer from life-threatening abnormal heart racing that originates from the lower chamber of the heart. These patients will often need an implantable defibrillator which has the ability to shock the heart back to a normal heart rhythm, but this does not prevent them from getting frequent recurrences of the bad heart rhythm needing shocks from the device. This can be painful and potentially harmful. Medicines to prevent recurrences of shocks are not very effective and have many side effects. An alternative to medicines for this is a procedure called a catheter ablation in which a wire is passed up through the blood vessels of the leg into the heart and used to find the short circuits which cause the dangerous heart rhythm. When the spot causing the trouble is found, the investigators can burn it ("ablate" it). This procedure is challenging and methods are needed to make it more effective and easier to do. One of the main ways for finding the short circuits involves using the electrocardiogram (the "ECG"). The regular ECG is simplistic and only makes use of recordings from 10 sites (6 precordial sites and 4 sites on both upper and lower limbs) on the body surface. The investigators are testing whether making recordings from 120 sites on the chest and back and using special computerized analysis of the recordings can help make catheter ablation for dangerous heart rhythms more effective.

DETAILED DESCRIPTION:
Several conventional and advanced mapping techniques are frequently utilized to accomplish a successful catheter ablation. Many of these mapping techniques (activation mapping, entrainment mapping) are hampered by either hemodynamic instability of some tachycardias or non-sustainability of others. Pacemapping is a commonly used tool for mapping non-sustained or hemodynamically unstable VT, which is based upon the principle that activation of the heart from a given site will yield a reproducible body surface electrocardiogram (ECG) morphology and that pacing from a site very close to the site at which VT activates the heart will result in a matching ECG morphology. This technique, however, is limited by imperfect accuracy and spatial resolution, subjectivity of interpretation leading to marked inter-observer variability in the perceived quality of a morphologic match, and by the need for an intuitive interpretation of the ECG to direct catheter manipulation. We hypothesize that one can improve the accuracy with which the origin of VT is localized by applying body surface potential mapping (BSPM), using data derived from 120 simultaneously acquired ECGs.

Objectives:

1. To quantify the similarity between BSPM waveforms during induced VT and during pacemapping or between two different pacing sites using two waveform comparison metrics, the correlation coefficient (CORR) and the root mean square error (RMSE) and to test the validity of these metrics as markers of proximity of the pacing site to the site of earliest ventricular activation.
2. To compare the accuracy with which the origin of ventricular tachycardia is localized via pacemapping by applying (BSPM), which uses data derived from 120 simultaneously acquired ECGs, to the accuracy of localization with different ECG subsets e.g. 12-lead ECG and X, Y and Z leads.

Patient and methods:

We anticipate that our patients will fall in one of the flowing 4 groups:

Group A:Patients with focal VT in structurally normal heart. Group B:Patients with scar related VT in which the exit site can be identified. Group C:Patients with scar related VT in which the exit site cannot be identified.Group D:Patients presenting with SVT.

For all groups, data for body-surface potential mapping (BSPM) will be recorded during induced VT (Group A& B), pacing from virtual VT exit sites which are several points selected around the scar margin to represent the VT exit site (group C) or index pacing site which is a pacing site selected as a reference in the RV of patients presented with SVT (group D) and from different pacemapping sites including successful and unsuccessful ablation sites if applicable. All data will be imported into customized software.

The improvement in the arithmetic value of the two comparison metrics will be tested as the site of pacing approaches the site of earliest ventricular activation (Groups A&B) or virtual VT exit sites in group C or the index pacing site (in group D). The best CORR and RMSE between the BSPM obtained during VT (in group A and B)/virtual VT exit sites (in group C) or index pacing site (group D) and different pacing sites (including successful and unsuccessful ablation sites) will be recorded. A simple linear regression will be used to compare the CORR and RMSE difference at each pacing site to distance between this pacing site and the successful ablation site as a surrogate of the best pace-match (in group A and B) or the corresponding virtual VT exit site (in group C) or index pacing site (group D). P value <0.05 will be considered significant. The mean sensitivity, specificity, and positive- and negative-predictive accuracies of the arithmetic metrics in determining the VT origin/exit site will be determined. We will repeat the previous protocol using different ECG subsets including 12 lead ECGs and X, Y and Z leads. The predictive accuracies for different subsets of electrodes will be measured and compared to those derived from using the whole BSPM obtained from the 120 ECG leads.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting with sustained monomorphic VT who are amenable to VT ablation.
* Patients referred for ablation of supraventricular tachycardia.

Exclusion Criteria:

* Patients presenting with ventricular tachycardia if no sustained tachycardia can be induced, or if in that particular patient pace-mapping is known to be an inaccurate method of mapping (e.g. in bundle branch reentry VT or fascicular VT).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from consecutive patients referred for ablation of sustained ventricular tachycardia with or without structural heart disease or Patients referred for ablation of supraventricular tachycardia to the QEII Health Sciences Centre, in Halifax, NS.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Correlating the arithmetic markers (CORR and MAD) to the distance between the pacing site and origin of the ventricular tachycardia or the index pacing site. | One year

CONTACTS AND LOCATIONS:
Overall Officials: John A Sapp, MD, FRCPC, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Capital District Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poole JE, Johnson GW, Hellkamp AS, Anderson J, Callans DJ, Raitt MH, Reddy RK, Marchlinski FE, Yee R, Guarnieri T, Talajic M, Wilber DJ, Fishbein DP, Packer DL, Mark DB, Lee KL, Bardy GH. Prognostic importance of defibrillator shocks in patients with heart failure. N Engl J Med. 2008 Sep 4;359(10):1009-17. doi: 10.1056/NEJMoa071098. PMID 18768944
- [Background] Aliot EM, Stevenson WG, Almendral-Garrote JM, Bogun F, Calkins CH, Delacretaz E, Della Bella P, Hindricks G, Jais P, Josephson ME, Kautzner J, Kay GN, Kuck KH, Lerman BB, Marchlinski F, Reddy V, Schalij MJ, Schilling R, Soejima K, Wilber D; European Heart Rhythm Association (EHRA); Registered Branch of the European Society of Cardiology (ESC); Heart Rhythm Society (HRS); American College of Cardiology (ACC); American Heart Association (AHA). EHRA/HRS Expert Consensus on Catheter Ablation of Ventricular Arrhythmias: developed in a partnership with the European Heart Rhythm Association (EHRA), a Registered Branch of the European Society of Cardiology (ESC), and the Heart Rhythm Society (HRS); in collaboration with the American College of Cardiology (ACC) and the American Heart Association (AHA). Heart Rhythm. 2009 Jun;6(6):886-933. doi: 10.1016/j.hrthm.2009.04.030. No abstract available. PMID 19467519
- [Background] Stevenson WG, Soejima K. Catheter ablation for ventricular tachycardia. Circulation. 2007 May 29;115(21):2750-60. doi: 10.1161/CIRCULATIONAHA.106.655720. No abstract available. PMID 17533195
- [Background] Stevenson WG. In: Wilber D, Packer DL, Stevenson WG, eds. Catheter Ablation of Cardiac Arrhythmias: Basic Concepts and clinical Application. 3rd Edition: Blackwell Publishing; 2008:315-324.
- [Background] Gerstenfeld EP, Dixit S, Callans DJ, Rajawat Y, Rho R, Marchlinski FE. Quantitative comparison of spontaneous and paced 12-lead electrocardiogram during right ventricular outflow tract ventricular tachycardia. J Am Coll Cardiol. 2003 Jun 4;41(11):2046-53. doi: 10.1016/s0735-1097(03)00427-3. PMID 12798580
- [Background] American College of Cardiology/American Heart Association Task Force on Clinical Data Standards (ACC/AHA/HRS Writing Committee to Develop Data Standards on Electrophysiology); Buxton AE, Calkins H, Callans DJ, DiMarco JP, Fisher JD, Greene HL, Haines DE, Hayes DL, Heidenreich PA, Miller JM, Poppas A, Prystowsky EN, Schoenfeld MH, Zimetbaum PJ, Goff DC, Grover FL, Malenka DJ, Peterson ED, Radford MJ, Redberg RF. ACC/AHA/HRS 2006 key data elements and definitions for electrophysiological studies and procedures: a report of the American College of Cardiology/American Heart Association Task Force on Clinical Data Standards (ACC/AHA/HRS Writing Committee to Develop Data Standards on Electrophysiology). Circulation. 2006 Dec 5;114(23):2534-70. doi: 10.1161/CIRCULATIONAHA.106.180199. Epub 2006 Nov 27. No abstract available. PMID 17130345
- [Background] Zipes DP, Camm AJ, Borggrefe M, Buxton AE, Chaitman B, Fromer M, Gregoratos G, Klein G, Moss AJ, Myerburg RJ, Priori SG, Quinones MA, Roden DM, Silka MJ, Tracy C, Smith SC, Jr., Jacobs AK, Adams CD, Antman EM, Anderson JL, Hunt SA, Halperin JL, Nishimura R, Ornato JP, Page RL, Riegel B, Blanc JJ, Budaj A, Dean V, Deckers JW, Despres C, Dickstein K, Lekakis J, McGregor K, Metra M, Morais J, Osterspey A, Tamargo JL, Zamorano JL. ACC/AHA/ESC 2006 Guidelines for Management of Patients With Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death: a report of the American College of Cardiology/American Heart Association Task Force and the European Society of Cardiology Committee for Practice Guidelines (writing committee to develop Guidelines for Management of Patients With Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death): developed in collaboration with the European Heart Rhythm Association and the Heart Rhythm Society. Circulation. 2006;114(10):e385-484.
- [Background] de Bakker JM, van Capelle FJ, Janse MJ, Tasseron S, Vermeulen JT, de Jonge N, Lahpor JR. Slow conduction in the infarcted human heart. 'Zigzag' course of activation. Circulation. 1993 Sep;88(3):915-26. doi: 10.1161/01.cir.88.3.915. PMID 8353918